CLINICAL TRIAL: NCT02657174
Title: Effectiveness of Low Level Laser at the Auriculotherapy Points, in Reducing Postoperative Pain in Third Molar Surgery
Brief Title: Evaluation of Low-level Laser at Auriculotherapy Points to Reduce Postoperative Pain in Inferior Third Molar Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Anna Carolina Ratto Tempestini Horliana, PhD, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1.100.869
Record Dates: First submitted 2016-01-11; First posted 2016-01-15 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Pain
Keywords: third molar; auriculotherapy; inflammation; pain
MeSH Terms: conditions — Pain; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- G1- experimental active comparator group (Experimental): G1 - (Experimental) 40 third molars surgeries will be performed in a conventional manner. At the end of surgery low level laser in auricular acupuncture points will be applied for prevention of inflammation and pain in a split-mouth design.
  Interventions: Device: low level laser in auricular acupuncture points
- G2- control group (Placebo Comparator): G2 - (Control) 40 third molars surgeries will be performed in the conventional manner, identically to the G1. At the end of surgery low level laser device off in auricular acupuncture points will be applied. The patient will receive low level laser with a protection of lead in the laser nozzle, in order to block the passage of light, in the same auricular points used in G1, with split-mouth design.
  Interventions: Device: low level laser device off in auricular acupuncture points

INTERVENTIONS:
Device: low level laser in auricular acupuncture points — 40 third molars surgeries will be performed in a conventional manner. At the end of surgery, low level laser will be applied at auricular points for prevention of inflammation and pain in the immediate post-operative period (baseline).The operator will mark the points that will be irradiated on the outer atrium of the patient with red gel pen to avoid interference with red laser (λ = 660 nm). The low level laser points will be irradiated in the same operated side.
  Arms: G1- experimental active comparator group
Device: low level laser device off in auricular acupuncture points — 40 surgeries will be performed in the conventional manner, identically to the G1. The patient will receive low level laser with a protection of lead in the laser nozzle, in order to block the passage of light, in the same auricular points used in G1.
  Arms: G2- control group

SUMMARY:
The association between low level laser and auricular acupuncture can be an alternative when conventional drugs are contraindicated or to reduce the quantity of these postoperative medications. The objective of this study is to evaluate the efficiency of low level laser at auriculotherapy points in reducing postoperative pain in lower third molar surgery. Eighty third molars surgeries will be performed in 40 healthy patients by a split-mouth design. Immediately after surgery, each side of the patient's mouth will be randomly treated with different regimens in a double-blind design: low level laser in auricular acupuncture points or simulation of its use. This treatment will be performed at 24 and 48 hours after surgery. The primary variable is the post-operative pain. The secondary variables are trismus, edema and local temperature. They will be assessed at baseline, 24 hours, 48 hours and seven days after surgery.The blood samples for analysis of systemic inflammatory cytokines (TNF-α, interleukin 1, interleukin 6 and interleukin 8) will be assessed at baseline and 24 hours after surgery.

DETAILED DESCRIPTION:
Third molar surgery is the most common surgical procedure in dentistry. A comfortable, fast postoperative return to daily activities has increased the need to control inflammation and its signs and symptoms, such as pain and edema. Anti-inflammatories and analgesics have been used for this purpose, but they are not exempt from adverse effects, such as allergies and chronic gastritis, not to mention the medicine costs. The association between low level laser and auricular acupuncture can be an alternative when conventional drugs are contraindicated or to reduce the quantity of these postoperative medications. Among the advantages, we can mention the low risk of side effects, low cost and simplicity of application. The objective of this study is to evaluate the efficiency of low level laser at auriculotherapy points in reducing postoperative pain in lower third molar surgery. Eighty bilateral, symmetrical lower third molars surgeries will be performed in 40 healthy patients. Each patient will be his or her own control, through a split-mouth technique. Immediately after surgery, each side of the patient's mouth will be randomly treated with different regimens in a double-blind design: low level laser in auricular acupuncture points or simulation of its use (contralateral side). This regimen will be repeated at 24 and 48 hours after surgery. All patients will receive the same medication (paracetamol) and will be oriented to take it only if they have pain. Neither the surgeon nor the patients know the assigned treatment. The primary variable is the post-operative pain assessed by visual analog scale, and the secondary variables are trismus, edema, local temperature. Dysphagia and presence of infection (systemic temperature, lymphadenopathy) will also be evaluated. These variables will be assessed at baseline, 24 hours, 48 hours and seven days after surgery. All adverse effects will be recorded. The blood samples for analysis of systemic inflammatory cytokines (TNF-α, interleukin 1, interleukin 6 and interleukin 8) will be assessed at baseline and 24 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* healthy patients (negative medical history)
* teeth in position II B according classification of Pell and Gregory
* third molar with extraction indication (recurrent infections, poor position, orthodontic indication) with professional statement in writing.

Exclusion Criteria:

* allergic to any drug used in the research (e.g.paracetamol)
* pregnant or breastfeeding women
* smokers
* patients submitted to radiotherapy in the head and neck, systemic or local infection (e.g., pericoronitis or periodontal abscess)
* patients with injuries or radiolucent images associated with the third molar
* patients who have used anti-inflammatory drugs in the last three months
* drug users
* patients who present any complications during surgery (e.g., bleeding, surgical difficulty, surgery longer than 90 minutes).

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-11 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Change in of post-operative pain by applying a visual analog scale | baseline
  The pain will be assessed by applying a visual analog scale, consisting of a 100-mm line numbered in centimeters, with two closed ends. One end is labeled "0" and the other "100", meaning no pain and terrible pain, respectively. Each patient will be instructed to mark a vertical line with the point that best matches the intensity of pain during the evaluation. Instructions on marking will always be given to the patient by the same operator.
Change in of post-operative pain by applying a visual analog scale | Postoperative period: 24 hours after surgery
  The pain will be assessed by applying a visual analog scale, consisting of a 100-mm line numbered in centimeters, with two closed ends. One end is labeled "0" and the other "100", meaning no pain and terrible pain, respectively. Each patient will be instructed to mark a vertical line with the point that best matches the intensity of pain during the evaluation. Instructions on marking will always be given to the patient by the same operator.
Change in of post-operative pain by applying a visual analog scale | Postoperative period: 48 hours after surgery
  The pain will be assessed by applying a visual analog scale, consisting of a 100-mm line numbered in centimeters, with two closed ends. One end is labeled "0" and the other "100", meaning no pain and terrible pain, respectively. Each patient will be instructed to mark a vertical line with the point that best matches the intensity of pain during the evaluation. Instructions on marking will always be given to the patient by the same operator.
Change in of post-operative pain by applying a visual analog scale | Postoperative period: 7 days after surgery
  The pain will be assessed by applying a visual analog scale, consisting of a 100-mm line numbered in centimeters, with two closed ends. One end is labeled "0" and the other "100", meaning no pain and terrible pain, respectively. Each patient will be instructed to mark a vertical line with the point that best matches the intensity of pain during the evaluation. Instructions on marking will always be given to the patient by the same operator.

SECONDARY OUTCOMES:
Changes in edema | baseline
  The criteria for the determination of edema will follow pre-established measurements: (I) Corner of the eye to angle of the jaw (II) Tragus to the labial commissure and (III) Tragus to pogonion.
Changes in mouth opening assessed by the inter-incisor measurement | baseline
  For evaluation of the presence of trismus the inter-incisor measurement (distance between the incisal edge of the maxillary central incisor and lower) will be used with a digital caliper. During clinical examination (one week before the surgery), the patient will be asked to perform his/her maximum mouth opening, which will be measured in millimeters.
Changes in local temperature | baseline
  The local temperature will be measured in the mandibular angle region 2 cm above the lower jaw board (Safety 1st® model "No Touch Forehead", Columbus, USA).
Changes in edema | Postoperative period: 24 hours after surgery
  The criteria for the determination of edema will follow pre-established measurements: (I) Corner of the eye to angle of the jaw (II) Tragus to the labial commissure and (III) Tragus to pogonion.
Changes in mouth opening assessed by the inter-incisor measurement | Postoperative period: 24 hours after surgery
  For evaluation of the presence of trismus the inter-incisor measurement (distance between the incisal edge of the maxillary central incisor and lower) will be used with a digital caliper. During clinical examination (one week before the surgery), the patient will be asked to perform his/her maximum mouth opening, which will be measured in millimeters.
Changes in local temperature | Postoperative period: 24 hours after surgery
  The local temperature will be measured in the mandibular angle region 2 cm above the lower jaw board (Safety 1st® model "No Touch Forehead", Columbus, USA).
Changes in edema | Postoperative period: 48 hours after surgery
  The criteria for the determination of edema will follow pre-established measurements: (I) Corner of the eye to angle of the jaw (II) Tragus to the labial commissure and (III) Tragus to pogonion.
Changes in mouth opening assessed by the inter-incisor measurement | Postoperative period: 48 hours after surgery
  For evaluation of the presence of trismus the inter-incisor measurement (distance between the incisal edge of the maxillary central incisor and lower) will be used with a digital caliper. During clinical examination (one week before the surgery), the patient will be asked to perform his/her maximum mouth opening, which will be measured in millimeters.
Changes in local temperature | Postoperative period: 48 hours after surgery
  The local temperature will be measured in the mandibular angle region 2 cm above the lower jaw board (Safety 1st® model "No Touch Forehead", Columbus, USA).
Changes in edema | Postoperative period: 7 days after surgery
  The criteria for the determination of edema will follow pre-established measurements: (I) Corner of the eye to angle of the jaw (II) Tragus to the labial commissure and (III) Tragus to pogonion.
Changes in mouth opening assessed by the inter-incisor measurement | Postoperative period: 7 days after surgery
  For evaluation of the presence of trismus the inter-incisor measurement (distance between the incisal edge of the maxillary central incisor and lower) will be used with a digital caliper. During clinical examination (one week before the surgery), the patient will be asked to perform his/her maximum mouth opening, which will be measured in millimeters.
Changes in local temperature | Postoperative period: 7 days after surgery
  The local temperature will be measured in the mandibular angle region 2 cm above the lower jaw board (Safety 1st® model "No Touch Forehead", Columbus, USA).

OTHER OUTCOMES:
Changes in systemic temperature | baseline
  Fever (systemic) is an indicator of infection. Because in case of infection pain is usually worse, it may become a bias. The temperature will be measured using a digital thermometer (Safety 1st® model "No Touch Forehead", Columbus, USA).
Changes in dysphagia through a numerical scale | baseline
  The assessment of dysphagia will be conducted through a numerical scale: 0 - indicates total absence of dysphagia; 1 - dysphagia for solid food; 2 - dysphagia for any food, liquid or solid.
Changes in systemic temperature | Postoperative period: 24 hours after surgery
  Fever (systemic) is an indicator of infection. Because in case of infection pain is usually worse, it may become a bias. The temperature will be measured using a digital thermometer (Safety 1st® model "No Touch Forehead", Columbus, USA).
Changes in dysphagia through a numerical scale | Postoperative period: 24 hours after surgery
  The assessment of dysphagia will be conducted through a numerical scale: 0 - indicates total absence of dysphagia; 1 - dysphagia for solid food; 2 - dysphagia for any food, liquid or solid.
Changes in systemic temperature | Postoperative period: 48 hours after surgery
  Fever (systemic) is an indicator of infection. Because in case of infection pain is usually worse, it may become a bias. The temperature will be measured using a digital thermometer (Safety 1st® model "No Touch Forehead", Columbus, USA).
Changes in dysphagia through a numerical scale | Postoperative period: 48 hours after surgery
  The assessment of dysphagia will be conducted through a numerical scale: 0 - indicates total absence of dysphagia; 1 - dysphagia for solid food; 2 - dysphagia for any food, liquid or solid.
Changes in systemic temperature | Postoperative period: 7 days after surgery
  Fever (systemic) is an indicator of infection. Because in case of infection pain is usually worse, it may become a bias. The temperature will be measured using a digital thermometer (Safety 1st® model "No Touch Forehead", Columbus, USA).
Changes in dysphagia through a numerical scale | Postoperative period: 7 days after surgery
  The assessment of dysphagia will be conducted through a numerical scale: 0 - indicates total absence of dysphagia; 1 - dysphagia for solid food; 2 - dysphagia for any food, liquid or solid.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Carolina RT Horliana, PhD, Principal Investigator — Nove de Julho University
Locations (1):
- Nove de Julho University (UNINOVE), São Paulo, Brazil

REFERENCES:
- [Derived] Sampaio-Filho H, Bussadori SK, Goncalves MLL, da Silva DFT, Borsatto MC, Tortamano IP, Longo PL, Pavani C, Fernandes KPS, Mesquita-Ferrari RA, Horliana ACRT. Low-level laser treatment applied at auriculotherapy points to reduce postoperative pain in third molar surgery: A randomized, controlled, single-blinded study. PLoS One. 2018 Jun 19;13(6):e0197989. doi: 10.1371/journal.pone.0197989. eCollection 2018. PMID 29920521
- [Derived] Sampaio-Filho H, Sotto-Ramos J, Pinto EH, Cabral MR, Longo PL, Tortamano IP, Marcos RL, Silva DF, Pavani C, Horliana AC. Evaluation of low-level laser at auriculotherapy points to reduce postoperative pain in inferior third molar surgery: study protocol for a randomized controlled trial. Trials. 2016 Sep 2;17(1):432. doi: 10.1186/s13063-016-1540-9. PMID 27590454